CLINICAL TRIAL: NCT01165749
Title: A Randomized Trial of Moderate Intensity Exercise Training in Patients With Hypertrophic Cardiomyopathy
Brief Title: Exercise Study Including Patients With Hypertrophic Cardiomyopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Dr. Euan Ashley MRCP, DPhil, Stanford University School of Medicine
Other Study IDs: SU-05062010-5902; 18518
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Cardiomyopathy, Hypertrophic
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: stop exercising

SUMMARY:
The long term health and cardiovascular benefits of a regular exercise program have been well-established. National guidelines recommend involvement in moderate aerobic fitness (i.e. walking, bicycling, light jogging, swimming) for patients with hypertrophic cardiomyopathy (HCM). However, data on potential benefits of recreational exercise, useful parameters for risk stratification, and methods of devising individual exercise prescriptions are completely lacking. The specific aims of this study are: 1) to devise a safe moderate intensity exercise training program in patients with HCM, and 2) to determine whether exercise training improves ability to perform activities and tasks, heart size and function, and quality of life in patients with HCM.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 - 80 years old.
2. Diagnosis of hypertrophic cardiomyopathy, defined by the presence of unexplained left-ventricular hypertrophy (wall thickening) > 13 mm in any wall segment.
3. Exercise £ 30 minutes, 1 day per week for the previous 3 months.
4. Agreement to be a participant in the study protocol and willing/able to return for follow-up.

Exclusion Criteria:

1. History of exercise-induced syncope or arrhythmias (ventricular tachycardia or non-sustained ventricular tachycardia).
2. Medically refractory LV outflow tract obstruction being evaluated for septal reduction therapy.
3. Less than 3 months post septal reduction therapy (surgery or catheter based intervention).
4. Hypotensive response to exercise (> 20 mmHg drop in systolic blood pressure from peak blood pressure to post exercise blood pressure).
5. Pregnancy.
6. ICD placement in last 3 months or scheduled.
7. Life expectancy less than 12 months.
8. Inability to exercise due to orthopedic or other non-cardiovascular limitations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with hypertrophic cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-12 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Improvement in ability to perform activities and tasks. | 4 months

SECONDARY OUTCOMES:
Improvement in heart size and function and quality of life (QOL). | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Euan Ashley MRCP, DPhil, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States